CLINICAL TRIAL: NCT04498195
Title: Effect of a Walking Intervention on Cognitive Function in Individuals With Mild Cognitive Impairment: A Knowledge Translation to Practice Pilot Project
Brief Title: Walking on Cognitive Function in Individuals With Mild Cognitive Impairment: A Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Merritt University (Other)
Responsible Party: Principal Investigator, Gasong Yun Nickerson, DNP graduate, Samuel Merritt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMUIRB#19-013
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Impairment, Mild
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increase physical activity and exercise (Experimental)
  Interventions: Behavioral: increased exercise and physical activity

INTERVENTIONS:
Behavioral: increased exercise and physical activity — Participants were encouraged to increase physical activity for 12-week study duration and wear an activity tracker for a minimum of 12 hours a day.

SUMMARY:
Background: Many studies suggest physical activity reduces risk of dementia and improves global cognitive function in individuals with mild cognitive impairment (MCI). Using commercial wearable technology to measure daily steps is feasible in this population.

Objectives: The purpose of this pilot study was to explore whether 12 weeks of increased physical activity improved cognitive function in individuals with MCI. A wearable activity tracker was used to measure participants' daily steps as a quantifiable measure of daily activity level.

Design: This was a one-group pretest-posttest study.

Setting: Established memory clinic patients within a neurology department in Northern California during 2019.

Participants: 17 enrolled and 14 included for data analysis. There were 7 females and 7 males whose mean age was 76.21 (SD 2.69). 12 participants were White, which reflected the clinic population.

Intervention: Participants were asked to wear an activity tracker for approximately 12 hours a day for 12 weeks and to increase their physical activity as much as possible. They were provided twice a month telephone support.

Measurements: The Montreal Cognitive Assessment (MoCA) was used to measure pretest-posttest cognitive function. Timed Up and Go (TUG) was used to assess fall risk at enrollment. Cumulative step count for the study period was measured with an activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Participants had a score of 0.5 on the Clinical Dementia Rating and are on a stable medication regimen for 3 months prior to enrollment.

Exclusion Criteria:

* a diagnosis of dementia; receiving chemotherapy; unstable chronic diseases; surgery with general anesthesia in the prior 3 months; MRI-confirmed brain damage from trauma, stroke, or other neurological disorder; a myocardial infarction < 1 year; a serious or non-healing wound, ulcer, or bone fracture; TUG ≥ 12 seconds; MoCA score >26 or <16; already using a wearable activity tracker; lacked access to the internet; or non-English speaking.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Whether increasing the number of daily steps among older adults with mild cognitive impairment would improve their cognitive functioning. | 12 weeks
  participants would wear an activity tracker and increase physical activity as much as possible within their comfort level. Participants will be tested for pretest MoCA for cognitive function and TUG for fall risk. After 12 weeks, participants will be tested for posttest MoCA to find any cognitive function change.

CONTACTS AND LOCATIONS:
Locations (1):
- Sutter Medical Neuroscience, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No